CLINICAL TRIAL: NCT00165334
Title: Phase II Trial of Cetuximab Plus Vinorelbine in Previously Untreated Patients > 70 With Advanced NSCLC
Brief Title: Cetuximab and Vinorelbine in Elderly Subjects With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-422
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Cetuximab; Vinorelbine; Navelbine; Previously untreated lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Vinorelbine

INTERVENTIONS:
Drug: Cetuximab
Drug: Vinorelbine (Navelbine)

SUMMARY:
The purpose of this study is it to determine how well patients with non-small cell lung cancer respond to cetuximab plus vinorelbine. We would also like to determine the safety of cetuximab plus vinorelbine in people 70 years of age or older with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
* Each cycle of study treatment is 21 days long. Cetuximab will be administered weekly intravenously on days 1, 8 and 15 of the 21-day cycle.
* Vinorelbine will be administered intravenously on days 1 and 8 of the 21-day cycle. On the days when the patient receives both cetuximab and vinorelbine, cetuximab will be given first.
* For the first cycle only, the first infusion of cetuximab will be in a larger dose and over a two-hour period of time. Beginning with the second treatment of cetuximab, the patient will receive a smaller dose over a one-hour period of time.
* For the first treatment of cetuximab, the patient will have their blood pressure, temperature, breathing rate and heart rate (vital signs) taken at the following time points: before the infusion, 1/2 hour into the infusion, at the end of infusion, and one hour after the infusion.
* For each subsequent cetuximab treatment, vital signs will be taken before each infusion and one hour after the end of infusion. The patient will be required to remain in the infusion room for one hour after the end of each cetuximab treatment for observation.
* CT scan(s), MRI(s), and/or x-rays(s) of the site(s) of cancer will be done every six weeks (every two cycles) while the patient is on the study to assess the extent of the cancer and the response to treatment.
* The duration of active participation in this study will depend on how the patients non-small cell lung cancer responds to treatment and how well they tolerate the treatment. The patient may receive up to six cycles of treatment with vinorelbine and cetuximab. After these six cycles the patient may continue on cetuximab alone as long as they are tolerating the drug and the cancer doesn't progress.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or greater
* Stage IV or IIIB Non-small cell lung cancer
* Must at least be able to walk and capable of taking care of yourself although unable to carry out work activities
* 3 or more weeks since completing prior radiotherapy
* 3 or more weeks since prior major surgery
* Blood tests that show your kidneys, liver and bone marrow to be working adequately
* Life expectancy of 8 weeks or more

Exclusion Criteria:

* Prior anticancer therapy within the past 3 years, including chemotherapy
* Other currently active cancer
* Uncontrolled Central Nervous System (CNS) problems
* Pre-existing disease or abnormality of the nervous system
* Hepatitis or Known HIV
* Active uncontrolled infection
* Incomplete healing from previous major surgery
* Significant history of uncontrolled cardiac disease such as high blood pressure, recent heart attack (within past 6 months), congestive heart failure, etc.
* Prior therapy which targets the ErbB pathway
* Prior severe infusion reaction to an antibody
* Chemotherapy or other investigational agent not indicated in the study protocol occuring at the same time as this study treatment
* A medical condition that could make it unsafe for you to participate in this study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine the overall response of cetuximab plus vinorelbine in patients 70 years or older with non-small lung cancer.

SECONDARY OUTCOMES:
To determine the safety of cetuximab plus vinorelbine in patients 70 years or older
to determine the time to progression and survival rates of patients treated with cetuximab plus vinorelbine.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Gridelli C, Perrone F, Gallo C, Cigolari S, Rossi A, Piantedosi F, Barbera S, Ferrau F, Piazza E, Rosetti F, Clerici M, Bertetto O, Robbiati SF, Frontini L, Sacco C, Castiglione F, Favaretto A, Novello S, Migliorino MR, Gasparini G, Galetta D, Iaffaioli RV, Gebbia V; MILES Investigators. Chemotherapy for elderly patients with advanced non-small-cell lung cancer: the Multicenter Italian Lung Cancer in the Elderly Study (MILES) phase III randomized trial. J Natl Cancer Inst. 2003 Mar 5;95(5):362-72. doi: 10.1093/jnci/95.5.362. PMID 12618501
- [Background] Effects of vinorelbine on quality of life and survival of elderly patients with advanced non-small-cell lung cancer. The Elderly Lung Cancer Vinorelbine Italian Study Group. J Natl Cancer Inst. 1999 Jan 6;91(1):66-72. doi: 10.1093/jnci/91.1.66. PMID 9890172